CLINICAL TRIAL: NCT04159103
Title: A Global, Phase 1/2, Open-Label, Dose Optimization Study to Evaluate the Safety, Pharmacodynamics, and Pharmacokinetics of mRNA-3927 in Participants With Propionic Acidemia
Brief Title: Open-Label Study of mRNA-3927 in Participants With Propionic Acidemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: mRNA-3927-P101; 2022-502910-10-00 (Other: Clinical Trials Information System (CTIS))
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Propionic Acidemia
Keywords: mRNA-3927; Propionic Aciduria; Metabolism, Inborn Errors; Genetic Diseases; Inborn Amino Acid Metabolism, Inborn Errors; Acidosis; Acid-Base Imbalance; Metabolic Diseases; Organic Acidemias; Moderna; mRNA
MeSH Terms: conditions — Propionic Acidemia; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Amino Acid Metabolism, Inborn Errors; Acidosis; Acid-Base Imbalance; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part 1 (Dose Optimization), Part 2 (Pivotal Study), and Part 3 (Infants) (Experimental): Part 1 (Dose Optimization): Participants (≥1 year of age) will receive single dose of mRNA-3927 by intravenous (IV) infusion every 2 weeks (Q2W) or every 3 weeks (Q3W) for up to 10 doses.
  Part 2 (Pivotal Study): Participants (≥1 year of age) will receive single dose of mRNA-3927 (identified during Dose Optimization Phase) by IV infusion Q2W for up to 26 doses or approximately 12 months. Part 3: Participants (<1 year of age) will receive single dose of mRNA-3927 (identified during Dose Optimization Phase) by IV infusion Q2W for up to 26 doses or approximately 12 months.
  Interventions: Biological: mRNA-3927

INTERVENTIONS:
Biological: mRNA-3927 — mRNA-3927 dispersion for IV infusion

SUMMARY:
This 3-part, Phase 1/2 study is designed to characterize the safety, tolerability, and pharmacological activity (as assessed by biomarker measurements) and to determine the selected dose of mRNA-3927 in participants with genetically confirmed propionic acidemia (PA). After establishing a dose with an acceptable safety and pharmacodynamic (PD) response for participants ≥1 year of age in Part 1, participants will be enrolled in Part 2 (which will serve as the pivotal study) to allow for determination of the efficacy, safety, and PD of mRNA-3927. Part 3 will evaluate the safety, efficacy and PD response of mRNA-3927 in infants (<1 year of age).

DETAILED DESCRIPTION:
During the Dose Optimization Stage, after each dose cohort is fully enrolled (≥1 year of age), and the dose-limiting toxicity (DLT) observation window of at least 14 days is complete for the final participant in that cohort, the Sponsor will review the totality of available safety data in conjunction with all available PK/PD data. Based on this review, the Sponsor will recommend a revised dose and/or dosing interval. The Sponsor will abide by predefined constraints as to the maximum percentage change in dose and dose interval. A maximum of 9 cohorts will be enrolled in Part 1 (Dose Optimization).

Upon establishment of a dose with an acceptable safety and PD activity in Part 1 (participants ≥1 year of age), additional participants will be enrolled into the study in Part 2 (participants ≥1 year of age) to allow for determination of the safety, efficacy, and PD of mRNA-3927. Part 3 will evaluate the safety, efficacy and PD response in infants (<1 year of age).

Participants in all the phases will participate in a predosing observational period, followed by a treatment period, and then a follow-up period after withdrawal of treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants ≥1 year of age are eligible to be included in the study only if all of the following criteria apply:

* ≥ 8 years of age at the time of consent/assent if enrolled as 1 of the first 2 participants in Part 1.
* ≥1 year of age at the time of consent/assent if enrolled after the first 2 participants in Part 1.
* Confirmed diagnosis of PA based on diagnosis by molecular genetic testing via central laboratory (PCCA and/or PCCB mutations).
* Part 2 only: At least one documented MDE in the 12-month period before consent.

Participants <1 Year of Age :

* Identification by newborn screening shortly after birth or having suspected PA by presenting with a spectrum of metabolic symptoms, and having a sibling diagnosed with PA. Participant may enter the Screening Period while awaiting genetic testing results, provided that all other eligibility criteria are met but would not be enrolled until diagnosis of PA is confirmed.
* For infants in the neonatal intensive care unit (NICU) only: ≥37 weeks gestational age at the time of birth without other conditions/comorbidities that in the opinion of the Investigator may interfere with the interpretation of study results.
* Body weight ≥3 kilograms (kg) at Screening.
* At least 1 documented PA-related event prior to Screening defined as the following criteria:

  * Clinical signs of metabolic deterioration consistent with PA (for example, vomiting, not feeding well/poor suck, heavy breathing, lethargy, absence of proper perfusion, abnormal movements including bicycling, abnormal tone, low body temperature, seizure[s]), OR
  * Meeting the criteria of MDE definition, OR
  * Evidence of laboratory abnormalities as evidenced by at least one of the following:
* Metabolic acidosis with elevated anion gap.
* Acute hyperammonemia.
* Neutropenia or thrombocytopenia.

Exclusion Criteria:

Participants of all ages are excluded from the study if during Screening any of the following criteria apply:

* Any individual with laboratory abnormalities considered to be clinically significant (for example, markedly out of range, associated with clinical symptoms) in the Investigator or Sponsor's opinion that could interfere with or limit the participation in the study.
* Estimated glomerular filtration rate (eGFR) <30 milliliters (mL)/minute/1.73 square meter (m^2) for participants of all ages receiving chronic dialysis.
* History of organ transplantation or planned organ transplantation during the period of study participation.
* Corrected QT interval (QTc) >480 milliseconds (ms) using Bazett's correction.
* Grade 3 or 4 heart failure according to the Modified Ross Heart Failure Classification for Children or the New York Heart Association Classification.
* Pregnant or breastfeeding.
* Other clinically significant conditions that in the Investigator's opinion could interfere with the safety of the participant, the interpretation of study results, or limit the participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Treatment-emergent Adverse Event (TEAE), Serious Adverse Events (SAE) and TEAEs Leading to Discontinuation | Day 1 (initial mRNA-3927 dose) up to Week 150 (End of Study)
Part 2: Change in Annualized Frequency of Clinical Event Committee (CEC)-adjudicated Metabolic Decompensation Events (MDEs) During 12-month Treatment Period With mRNA-3927 Compared to Annualized Frequency of CEC-adjudicated MDE During Pretreatment Period | Pretreatment period (12 months before consent to first mRNA-3927 dose in the study) up to Month 12
Part 3: Number of Participants with TEAEs, SAEs, Adverse Events (AEs) of Special Interest (AESIs) and TEAEs Leading to Discontinuation | Day 1 up to Week 73

SECONDARY OUTCOMES:
Part 1: Change From Baseline in Plasma 2-Methylcitrate (2-MC) and 3-Hydroxypropionic Acid (3-HP) Levels After Single and Repeated Administrations of mRNA-3927 | Baseline up to Week 40
  Baseline (predose levels) to postdose levels measured after single and after repeated administrations of mRNA-3927
Part 1: Maximum Observed Effect (Emax) of 2-MC and 3-HP After Single and Repeated Administrations of mRNA-3927 | Baseline up to Week 40
  Baseline (predose levels) to postdose levels measured after single and after repeated administrations of mRNA-3927
Part 1: Area Under the Effect Versus Time Curve (AUEC) of 2-MC and 3-HP After Single and Repeated Administrations of mRNA-3927 | Baseline up to Week 40
  Baseline (predose levels) to postdose levels measured after single and after repeated administrations of mRNA-3927
Part 1: Duration of Response (DOR) After Single and Repeated Administrations of mRNA-3927 | Baseline up to Week 40
  Baseline (predose levels) to postdose levels measured after single and after repeated administrations of mRNA-3927
Part 1: Maximum Observed Concentration (Cmax) of Propionyl-CoA Carboxylase Subunit α (PCCA) and Propionyl-CoA Carboxylase Subunit β (PCCB) mRNAs | Baseline up to Week 40
  Baseline (predose levels) to postdose levels measured after single and after repeated administrations of mRNA-3927
Part 1: Time of Cmax (Tmax) of PCCA and PCCB mRNAs | Baseline up to Week 40
  Baseline (predose levels) to postdose levels measured after single and after repeated administrations of mRNA-3927
Part 1: Area Under the Plasma Concentration-Time Curve (AUC) of PCCA and PCCB mRNAs | Baseline up to Week 40
  Baseline (predose levels) to postdose levels measured after single and after repeated administrations of mRNA-3927
Part 1: SM-86 Concentration After Single and Repeated Administrations of mRNA-3927 | Baseline up to Week 40
  Baseline (predose levels) to postdose levels measured after single and after repeated administrations of mRNA-3927
Part 1: Frequency of Anti-Polyethylene Glycol and Anti-Propionyl-CoA Carboxylase Antibodies | Day 1 (initial mRNA-3927 dose) up to Week 150 (End of Study)
Part 2: Change in Annualized Frequency of CEC-adjudicated MDE-related Hospitalizations During the 12-month Treatment Period With mRNA-3927 Compared to the Annualized Frequency of CEC-adjudicated MDE-related Hospitalizations During the Pretreatment Period | Pretreatment period (12 months before consent to first mRNA-3927 dose in the study) up to Month 12
Part 2: Change in Annualized Frequency of CEC-adjudicated PA-related Hospitalizations During the 12-month Treatment Period With mRNA-3927 Compared to the Annualized Frequency of CEC-adjudicated PA-related Hospitalizations During the Pretreatment Period | Pretreatment period (12 months before consent to first mRNA-3927 dose in the study) up to Month 12
Part 2: Change in Annualized Frequency of CEC-adjudicated MDEs During 12-month Treatment Period With mRNA-3927 Compared to Annualized Frequency of CEC-adjudicated MDE During Pretreatment Period by the Following Severity Grades: Grade 1, Grade 2, Grade 3 | Pretreatment period (12 months before consent to first mRNA-3927 dose in the study) up to Month 12
Parts 2 and 3: Change from Baseline in Pediatric Quality of Life Inventory (PedsQL) Total Score and Physical Function Score | Baseline up to Week 52
Parts 2 and 3: Change from Baseline in Methylmalonic Acidemia and Propionic Acidemia Questionnaire - Proximal Signs and Symptoms (MMAPAQ-PSS) Total Score | Baseline up to Week 52
Parts 2 and 3: Percentage of Participants Distributed into 'Mild', 'Moderate', and 'Severe' Categories Based on Investigator Global Assessment of Severity (IGA-S) Severity Levels | Baseline up to Week 52
Parts 2 and 3: Percentage of Participants Meeting 'Modestly Improved' or 'Much Improved' in Investigator Global Assessment of Improvement (IGA-I) | Baseline up to Week 52
Part 2: Change in Annualized Frequency of CEC-adjudicated PA-related Urgent Healthcare Encounters During 12-month Treatment Period Compared to Annualized Frequency of CEC-adjudicated PA-related Urgent Healthcare Encounters During Pretreatment Period | Pretreatment period (12 months before consent to first mRNA-3927 dose in the study) up to Month 12
Parts 2 and 3: Change From Baseline in Plasma 2-MC and 3-HP Levels After Administration of mRNA-3927 | Baseline up to Week 52
Parts 2 and 3: Area That is Below the Baseline and Above the Response Curve (AUC_Below_B) of 2-MC and 3-HP After Administration of mRNA-3927 | Baseline up to Week 52
Parts 2 and 3: Area Under the Curve That is AUC_Above_B - AUC_Below_B (AUC_Net_B) of 2-MC and 3-HP After Administration of mRNA-3927 | Baseline up to Week 52
Parts 2 and 3: Emax of 2-MC and 3-HP After Administration of mRNA-3927 | Baseline up to Week 52
Part 2: Number of Participants with TEAEs, SAEs, AESIs, and TEAEs Leading to Discontinuation | Day 1 up to Week 73
Part 3: Annualized Frequency of CEC-adjudicated MDEs | Baseline up to Week 52
Part 3: Annualized Frequency of CEC-adjudicated MDE-related Hospitalizations | Baseline up to Week 52
Part 3: Annualized Frequency of CEC-adjudicated PA-related Hospitalizations | Baseline up to Week 52
Part 3: Annualized Frequency of CEC-adjudicated MDEs by the Following MDE Severity Grades: Grade 1, Grade 2, Grade 3 | Baseline up to Week 52
Part 3: Annualized Frequency of CEC-adjudicated PA-related Urgent Healthcare Encounters | Baseline up to Week 52
Part 3: Cmax of PCCA and PCCB mRNAs | Baseline up to Week 52
Part 3: Tmax of PCCA and PCCB mRNAs | Baseline up to Week 52
Part 3: AUC of PCCA and PCCB mRNAs | Baseline up to Week 52
Part 3: Cmax of SM-86 and OL-56 | Baseline up to Week 52
Part 3: Tmax of SM-86 and OL-56 | Baseline up to Week 52
Part 3: AUC of SM-86 and OL-56 | Baseline up to Week 52

CONTACTS AND LOCATIONS:
Locations (35):
- United States (15):
  - UCSD Altman Clinical and Transalational Research Institute Building, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford, Stanford, California
  - Nicklaus Children's Hospital, Miami, Florida
  - University of South Florida - 12901 Bruce B Downs, Tampa, Florida
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Adult Outpatient Clinical Research Unit, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Hospitals, Ann Arbor, Michigan
  - Icahn School of Medicine at Mount Sinai - Clinical Research Unit, New York, New York
  - Duke University Medical System (Duke Health), Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center - 11100 Euclid Ave, Cleveland, Ohio
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
- Canada (2):
  - Stollery Children's Hospital University of Alberta, Edmonton, Alberta
  - Hospital For Sick Children, Toronto, Ontario
- France (2):
  - CHU de Marseille - Hôpital de la Timone, Marseille
  - Hôpital Necker - Enfants Malades, Paris
- Japan (3):
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - National Center for Child Health and Development, Tokyo
- Netherlands (2):
  - Erasmus MC, Rotterdam, South Holland
  - Universitair Medisch Centrum Utrecht - PPDS, Utrecht
- Saudi Arabia (3):
  - King Faisal Specialist Hospital & Research Center - Riyadh, Riyadh, Ar Riya
  - King Fahad Medical City, Riyadh, Ar Riya
  - King Abdullah Children's Specialist Hospital, Riyadh, Ar Riya
- Spain (4):
  - Hospital Sant Joan de Deu - PIN, Esplugues de Llobregat, Barcelona
  - Hospital Universitario Cruces, Barakaldo, Biscay
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
- United Kingdom (4):
  - University Hospital Birmingham NHS Foundation Trust, Birmingham
  - Birmingham Children's Hospital, Birmingham
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Willink Biochemical Genetics Unit - PPDS, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Attarwala H, Lumley M, Liang M, Ivaturi V, Senn J. Translational Pharmacokinetic/Pharmacodynamic Model for mRNA-3927, an Investigational Therapeutic for the Treatment of Propionic Acidemia. Nucleic Acid Ther. 2023 Apr;33(2):141-147. doi: 10.1089/nat.2022.0036. Epub 2022 Dec 27. PMID 36577040